CLINICAL TRIAL: NCT06678724
Title: Establishment of a Microfluidic Based Liquid Biopsy Platform for Recurrent/Metastatic Head and Neck Cancers Prognostication Using NK Cell IFN-γ Expression and CTM Correlation With DS-SACA Chip
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital Hsin-Chu Branch (Other); National Taiwan University Hospital, Yun-Lin Branch (Other)
Responsible Party: Sponsor
Other Study IDs: 202409056RINC
Record Dates: First submitted 2024-10-31; First posted 2024-11-07 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-10

CONDITIONS: Head and Neck Cancers- Squamous Cell; Head and Neck Cancer Metastatic; Recurrent Head and Neck Squamous Cell Carcinoma
Keywords: head and neck cancer; circulating tumor cell; CTC; circulating tumor emboli; CTM; NK cell; nature killer cell; prognosis; INF-gamma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Recurrent/Metastatic squamous cell carcinoma of the head and neck: Patient inclusion criteria, must fulfill with all the items below
  1. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0-2.>=20 years old.
  3. had pathologically confirmed squamous cell carcinoma of the oropharynx, oral cavity, hypopharynx, or larynx that was recurrent or metastatic and not curable by local therapy.
  4. had at least one tumor lesion measurable per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 5. Medical records during treatment are available.

SUMMARY:
The goal of this observational study is to learn about the prognostic value of circulation tumor emboli (CTM) in recurrent/metastatic head and neck cancer patients and also the changes of tumor microenvironment by different treatment modalities and drugs. The main questions it aims to answer are:

1. Investigators plan to correlate circulating tumor cells (CTC), circulating tumor emboli (CTM), and the composition of NK cells in CTM with clinical outcomes and establish their association with patient prognosis.
2. Investigators plan to understand the composition of NK cells and the immune cell components within CTM, and correlate these findings with treatment efficacy.

Patients with recurrent/metastatic head and neck cancer will be included after informed consent and investigators will collect blood samples for analysis from them under the treatment provided by their primary care physicians.

DETAILED DESCRIPTION:
Head and neck cancer, including oral, oropharyngeal and hypopharyngeal cancer, is the third most common type of cancer and the fourth leading cause of death of cancer among male patients in Taiwan according to the 2021 cancer registry. Despite surgery and adjuvant concurrent chemoradiotherapy (CCRT) for locally advanced head and neck cancer, there still were 20 to 30 % of patients who had recurrent disease within 2 years. For patients who were not suitable to receive surgery, the progression free survival was even worse, especially for those with HPV negative cancer In Taiwan, there is a special category of head and neck cancer which is associated with betel nut use and the molecular basis of this type of cancer is different. This is the most important reason why studies should be done in Taiwanese population.

In recent years, numbers of studies have confirmed that circulating tumor cells (CTCs) play a key role in the process of tumor metastasis and recurrence. The collection and analysis of CTCs is expected to provide patients with important information that was not easily available in the past and assist in planning of follow-up treatments strategy. However, CTCs research still faces many challenges, including: (1) The current clinical CTCs detection platform cannot tell whether the isolated cells contain the CTCs cluster or CTM from patient's liquid biopsy; (2) Lack of analytical technology to identify metastasis risk from the isolated CTCs and (3) how to analyze the immune microenvironment in CTM and apply it to formulate therapeutic strategy of the follow-up treatment.

As mentioned above, there are a group of patients who would experience recurrence locally or distant metastases within a short period of time after curative treatment. First, investigators want to establish a platform to predict recurrence and prognosis. By using the number of circulating tumor cells (CTCs), circulating tumor emboli (CTM) and INF-γ level incorporated with clinical factors to correlate with patient prognosis. Second, investigators want to evaluate the component of NK cells in CTM, and elucidate their correlation with different risk factors, including HPV status, smoking and betel nut use, treatment modalities, treatment drugs and patient prognosis.

This research will elucidate not only prognostic value of CTM, but also the changes of tumor microenvironment by different treatment modalities and drugs.

ELIGIBILITY:
Inclusion Criteria: must fulfill with all the items below

* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0-2.
* >=20 years old.
* had pathologically confirmed squamous cell carcinoma of the oropharynx, oral cavity, hypopharynx, or larynx that was recurrent or metastatic and not curable by local therapy.
* had at least one tumor lesion measurable per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Medical records during treatment are available.

Exclusion Criteria:

* Medical records during treatment unavailable
* Could not cooperate with blood sampling
* Without informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recurrent/Metastatic squamous cell carcinoma of the head and neck
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From enrollment to until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  The time from diagnosis as non-curable disease to clinically (physical examination or radiographically) confirmed disease progression or death from any cause, whichever came first.

SECONDARY OUTCOMES:
Overall survival (OS) | From date of enrollment until the date of death from any cause, whichever came first, assessed up to 60 months
  The time from diagnosis as non-curable disease to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University HsinChu Branch, Zhubei, HsinChu County, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: starting 6 months after publication